CLINICAL TRIAL: NCT05930444
Title: Multimodal Machine Learning for Auxiliary Diagnosis of Eye Diseases Using ChatGPT-based Natural Language Processing and Image Processing Techniques
Brief Title: Multimodal Machine Learning for Auxiliary Diagnosis of Eye Diseases
Status: Completed | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: The Affiliated Eye Hospital of Nanjing Medical University (Unknown); Suqian First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FD-EENT-20230625
Record Dates: First submitted 2023-06-25; First posted 2023-07-05 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Normal participants: Healthy individuals who have no concerns related to their eyes.
- Patients with Eye-related Chief Complaints: Individuals who have specific concerns or issues related to their eyes, which they consider as the main reason for seeking medical attention or making a complaint.
  Interventions: Diagnostic Test: Multimodal Machine Learning Program for Auxiliary Diagnosis of Eye Diseases

INTERVENTIONS:
Diagnostic Test: Multimodal Machine Learning Program for Auxiliary Diagnosis of Eye Diseases — Patients presenting with eye-related chief complaints initially complete a mobile phone application. This application utilizes patient medical history and relevant images (such as selfies and photos from eye examinations) to provide intelligent diagnosis. The diagnosis remains undisclosed to the patients. Subsequently, patients seek medical attention and undergo clinical examination by a skilled clinician. The clinical diagnosis is subsequently reviewed by a second experienced clinician. If the diagnoses align, it is considered the gold standard. In cases of discrepancy, the consensus reached by the two clinicians becomes the gold standard.
  Groups: Patients with Eye-related Chief Complaints

SUMMARY:
With rapid advancements in natural language processing and image processing, there is a growing potential for intelligent diagnosis utilizing chatGPT trained through high-quality ophthalmic consultation. Furthermore, by incorporating patient selfies, eye examination photos, and other image analysis techniques, the diagnostic capabilities can be further enhanced. The multi-center study aims to develop an auxiliary diagnostic program for eye diseases using multimodal machine learning techniques and evaluate its diagnostic efficacy in real-world outpatient clinics.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained;
* Participants should be able to have Chinese as their mother tongue, and be sufficiently able to read, write and understand Chinese;
* For normal participants: individuals should have no concerns related to their eyes.
* For participants with eye-related chief complaints: individuals should have specific concerns or issues related to their eyes.

Exclusion Criteria:

* Incomplete clinical data to support final diagnosis;
* Patients who, in the opinion of the attending physician or clinical study staff, are too medically unstable to participate in the study safely.

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The "normal participants" refers to individuals with no concerns or issues related to their eyes.
  The "participants with eye-related chief complaints" refers to patients from various eye clinics across China. Each participant must undergo comprehensive medical tests and have their medical records reviewed for diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 9825 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of multimodal machine learning program | from July 2023 to March 2024
  For each patient, the diagnoses generated by the multimodal machine learning program and the clinical diagnosis provided by skilled clinicians were documented and compared. Consistency between the two diagnoses indicates the program's precision in clinical practice.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Affiliated Eye Hospital of Nanjing Medical University, Nanjing
  - Fudan Eye & ENT Hospital, Shanghai
  - Suqian First People's Hospital, Suqian

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: The protocol has been published on 08 December 2023.
URL: https://pubmed.ncbi.nlm.nih.gov/38145231/

REFERENCES:
- [Derived] Ma R, Cheng Q, Yao J, Peng Z, Yan M, Lu J, Liao J, Tian L, Shu W, Zhang Y, Wang J, Jiang P, Xia W, Li X, Gan L, Zhao Y, Zhu J, Qin B, Jiang Q, Wang X, Lin X, Chen H, Zhu W, Xiang D, Nie B, Wang J, Guo J, Xue K, Cui H, Cheng J, Zhu X, Hong J, Shi F, Zhang R, Chen X, Zhao C. Multimodal machine learning enables AI chatbot to diagnose ophthalmic diseases and provide high-quality medical responses. NPJ Digit Med. 2025 Jan 27;8(1):64. doi: 10.1038/s41746-025-01461-0. PMID 39870855
- [Derived] Peng Z, Ma R, Zhang Y, Yan M, Lu J, Cheng Q, Liao J, Zhang Y, Wang J, Zhao Y, Zhu J, Qin B, Jiang Q, Shi F, Qian J, Chen X, Zhao C. Development and evaluation of multimodal AI for diagnosis and triage of ophthalmic diseases using ChatGPT and anterior segment images: protocol for a two-stage cross-sectional study. Front Artif Intell. 2023 Dec 8;6:1323924. doi: 10.3389/frai.2023.1323924. eCollection 2023. PMID 38145231
- See also: Development and evaluation of multimodal AI for diagnosis and triage of ophthalmic diseases using ChatGPT and anterior segment images: protocol for a two-stage cross-sectional study — https://pubmed.ncbi.nlm.nih.gov/38145231/